CLINICAL TRIAL: NCT06872762
Title: Does Heat Stress Improve the Acute Metabolic and Cardiovascular Adaptations to Exercise
Brief Title: Effect of Exercise and Heat Stress on Acute Cardiometabolic Adaptations in Healthy Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Travis Gibbons, Assistant Professor, Northern Arizona University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2224584
Record Dates: First submitted 2025-02-24; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Exercise; Heat Strain; Control Condition
Keywords: exercise; heat strain; glucose tolerance test; arterial compliance
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Random order, repeated measures, cross-over
Who Masked: Investigator
Masking Description: Researchers will be masked to data during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise (Experimental): Participants exercise for 90 minutes trying to remain cool with fans and limited clothing.
  Interventions: Behavioral: Exercise; Behavioral: Heat strain
- Heat strain (Experimental): Participants exercise for 90 minutes wearing winter and rain clothes to develop heat strain.
  Interventions: Behavioral: Exercise; Behavioral: Heat strain
- Control (Placebo Comparator): Resting control for 90 minutes. Not allowed to exercise.
  Interventions: Behavioral: Exercise; Behavioral: Heat strain

INTERVENTIONS:
Behavioral: Exercise — Exercise for 90 minutes (cycling) while minimizing thermal strain
Behavioral: Heat strain — Exercise for 90 minutes (cycling) while maximizing thermal strain

SUMMARY:
Life in space is completely void of physical and environmental stress. It is well known that living things need regular physical stress (e.g. exercise) to remain strong, functional and healthy. More and more research is showing that regular environmental stress, for example heat and hypoxia, can further improve physical health. Astronauts aboard the international space station (ISS) exercise for 1-2 hours every day to avoid physical deconditioning that would otherwise cause them to age rapidly in space. Although physical exercise is very effective in remedying this deconditioning, today's astronauts still have physiological changes that indicate accelerated aging. This is a cause for concern given NASA's priority to travel to mars within the next decade; a mission that will require at least double the duration in space for our astronauts. The investigators think that the complete absence of environmental stress, i.e., heat, may be contributing to the accelerated aging that occurs during spaceflight. Our study will assess the health effects of adding heat stress to exercise that could be performed in space by astronauts. The goal is to inform best practice for astronauts to avoid physical deconditioning during long-duration spaceflight. This information will also be relevant to life on earth as spaceflight is a model of inactivity here on earth. Therefore, the potential benefits of adding heat stress will likely translate to life in space and on earth.

DETAILED DESCRIPTION:
Experimental procedures:

Participants will visit the lab on seven occasions. Participants will be required to practice regular exercise and dietary habits that can be easily replicated in the 24 hours prior to every laboratory visit. Exercise and dietary patterns will be documented during the first visit and thereafter the participants will be reminded of these practices and instructed to match them as closely as possible in the 24 hours leading up to all subsequent visits. Participants will only be instructed to avoid heavy exercise in the 12 hours prior to testing sessions. On the first visit, participants will be introduced into the lab, where the investigators will give oral and written instruction detailing the procedures and associated risks related to participating. Details of the experimental visits are outlined below:

Familiarization Visit (1 hour):

* Familiarization and fitness test
* Lactate threshold and maximal aerobic power test on an upright cycle ergometer.

Experimental visit #1 (6 hours):

* Control exercise, heated exercise or control rest
* Rectal or esophageal thermistor will be inserted.
* Venous cannula will be inserted by trained phlebotomist (Chloe Gustafson, Dr Travis Gibbons).
* Cycling exercise for 90 minutes at 90% of lactate threshold with 2 pedestal fans to maximize heat loss and prevent core temperature increase to <1 ̊ C.
* 2.5 hours of resting recovery in semi-supine position.
* Vascular assessment.
* Glucose tolerance test (blood will be sampled for glucose and insulin 15, 30, 60 and 120 minutes after consuming a mixed macronutrient meal)
* Rectal thermistor and venous cannula will be removed and participant will leave.

Experimental visit #2 (6 hours):

* Control exercise, heated exercise or control rest
* Complete identical procedures as experimental visit #2 with the following exceptions:
* Cycling exercise for 90 minutes at 90% of lactate threshold.
* No fans will be used to maximal heat gain.
* Participants will wear a water impermeable jacket, pants and gloves, and wear a winter hat (beanie).
* Core temperature will be allowed to rise naturally but exercise will stop if core temperature reaches 40 ̊ C.

Experimental visit #3 (6 hours):

* Control exercise, heated exercise or control rest
* Complete identical procedures as experimental visit #2 with the following exceptions:
* Participant will rest comfortably in the semi-supine position for 90 minutes.

Follow-up assessments after experimental visits 1, 2, and 3 (1 hour):

* Rectal or esophageal thermistor will be inserted.
* Participant will lie comfortably for 10 minutes.
* Arterial stiffness assessment will be performed (3 minutes)
* A venous blood sample will be collected.
* Participant will complete 5-minute blood volume assessment via carbon monoxide rebreathing technique.
* A final blood draw will be performed.

ELIGIBILITY:
Inclusion Criteria:

-regularly physically active as determined via ParQ+

Exclusion Criteria:

* smokers
* bronchial asthma
* chronic obstructive pulmonary disease
* obese
* alcoholism
* requiring daily medications that may effect responses to exercise,
* anti-arrhythmogenics
* inhalers
* history of cardiovascular, respiratory, neurological, skeletal muscle disease
* irregular/absent menstrual cycle (females)
* unexpected responses to pre-experimental exercise tests
* previous diagnosis of heat stroke

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | 2 hours after intervention complete
  Glucose to insulin concentration ratio in serum.

SECONDARY OUTCOMES:
Arterial compliance | 2 hours after intervention complete
  Change in artery diameter (millimeter) assessed via ultrasound per change in artery pressure (mm Hg) assessed via tonometry.
Plasma volume expansion | 24 hours after intervention
  Plasma volume change measured with carbon monoxide rebreathe

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
I am concerned for privacy protection of our participants.